CLINICAL TRIAL: NCT01017029
Title: Early vs. Delayed EVERolimus in de Novo HEART Transplant Recipients: Optimization of the Safety/Efficacy Profile (EVERHEART Study)
Brief Title: Everolimus in de Novo Heart Transplant Recipients
Acronym: EVERHEART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001AIT16; 2009-011008-43
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Results first posted 2014-12-18 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2014-12

CONDITIONS: Cardiac Transplantation
MeSH Terms: interventions — Everolimus; Mycophenolic Acid

ARMS (2):
- Immediate introduction of everolimus (Active Comparator)
  Interventions: Drug: Everolimus
- Delayed introduction of everolimus (Experimental): delayed introduction) + Cyclosporin + steroids
  Interventions: Drug: Mycophenolate mofetil + Everolimus

INTERVENTIONS:
Drug: Everolimus
  Arms: Immediate introduction of everolimus
Drug: Mycophenolate mofetil + Everolimus
  Arms: Delayed introduction of everolimus

SUMMARY:
The purpose of this study, in de novo heart transplant patients, is to evaluate whether delayed introduction of everolimus reduces the occurrence of wound healing problems, pericardial and/or pleural effusion and early acute renal insufficiency, as compared with immediate introduction of everolimus, in the firs six months after heart transplantation.

ELIGIBILITY:
Inclusion criteria:

* Male or female cardiac transplant candidates 18-65 years of age undergoing primary heart transplantation.
* Glomerular filtration rate (GFR by MDRD) ≥ 40 mL/min/1.73 m2 at randomization

Exclusion criteria:

* Patients who are recipients of multiple solid organ transplants
* Patients who are HIV-positive or Hepatitis C positive (PCR only) or B-surface antigen positive;
* Presence of Donor/Recipients serological mismatch for Hepatitis B or C;
* Recipients of organ from donors positive for Hepatitis B-surface antigen;
* Panel Reactive Antibodies (cytotoxicity method) > 30%.
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2009-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- Italy (12):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Napoli

REFERENCES:
- [Derived] Potena L, Pellegrini C, Grigioni F, Amarelli C, Livi U, Maccherini M, Masciocco G, Faggian G, Lilla Della Monica P, Gerosa G, Marraudino N, Corda M, Boffini M; EVERHEART Investigators. Optimizing the Safety Profile of Everolimus by Delayed Initiation in De Novo Heart Transplant Recipients: Results of the Prospective Randomized Study EVERHEART. Transplantation. 2018 Mar;102(3):493-501. doi: 10.1097/TP.0000000000001945. PMID 28930797

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Introduction of Everolimus: Everolimus within 144 hours (5 days) after graft reperfusion + cyclosporine microemulsion + steroids
- Delayed Introduction of Everolimus: Mycophenolate mofetil (MMF) within 144 hours (5 days) after graft reperfusion + cyclosporine microemulsion + steroids. After 4 to 6 weeks since transplant, everolimus in place of MMF and dose of cyclosporine reduced.
Period: Overall Study
Arm/Group | Immediate Introduction of Everolimus | Delayed Introduction of Everolimus
Started | 89 | 92
Completed | 85 | 90
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Administrative problem | 0 | 1
Not completed — Death | 3 | 1

BASELINE CHARACTERISTICS:
Population: safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Introduction of Everolimus | Delayed Introduction of Everolimus | Total
Number analyzed (Participants) | 89 | 92 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.69 (10.15) | 52.95 (10.19) | 52.82 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 37
  Male | 73 | 71 | 144
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 88 | 88 | 176
  Black | 0 | 1 | 1
  Other | 1 | 3 | 4
Weight [Mean (Standard Deviation); unit: kilograms] | 74.38 (12.50) | 71.18 (12.75) | 72.76 (12.70)
Height [Mean (Standard Deviation); unit: centimeters] | 170.80 (7.69) | 170.10 (8.03) | 170.44 (7.85)
Calculated BMI [Mean (Standard Deviation); unit: kg/m2*] — Body Mass Index (BMI) Body mass divided by the square of their height.
  kg/m2* | 25.44 (3.65) | 24.48 (3.33) | 24.95 (3.52)

OUTCOME MEASURES:

1. Primary Outcome: Participants With at Least One Occurrence of Safety Composite Endpoint After 6 Months by Treatment Group
Description: Comparison of 6-month cumulative incidence of safety composite endpoint (wound healing delay) related to initial transplant surgery, pleural/pericardial effusions and occurrence of acute renal insufficiency, defined as estimated glomerular filtration rate (eGFR) ≤ 30 mL/min/1.73 m2, between delayed everolimus arm and immediate everolimus arm
Time Frame: 6 months
Population: safety population
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Immediate Introduction of Everolimus | Delayed Introduction of Everolimus
Number analyzed (Participants) | 89 | 92
participants | 40 [34.60 to 55.30] | 30 [23.00 to 42.20]
Statistical Analysis 1: Comparison: Immediate Introduction of Everolimus vs Delayed Introduction of Everolimus; Test type: Superiority or Other; p = 0.1043, Regression, Cox; Hazard Ratio (HR) = 1.482, 95% CI 2-sided [0.922 to 2.383]

2. Secondary Outcome: Partcipants With at Least One Occurrence of Each Safety Composite Endpoint Event After 6 Months by Treatment Group
Time Frame: 6 months
Population: safety population
Measure: Number (95% Confidence Interval); unit: participants
Units Other Than Participants: participants
Arm/Group | Immediate Introduction of Everolimus | Delayed Introduction of Everolimus
Number analyzed (Participants) | 89 | 92
participants
  Wound healing complication | 10 [4.7 to 17.8] | 8 [2.9 to 14.50]
  Pleural effusion | 1 [0.00 to 3.30] | 1 [0.00 to 3.20]
  Pericardial effusion | 30 [23.90 to 43.50] | 18 [11.50 to 27.70]
  eGFR ≤ 30 mL/min/1.73 m2 | 7 [2.30 to 13.50] | 8 [2.90 to 14.50]

3. Secondary Outcome: Hazard Cox's Model Analysis of Pericardial/Pleural Effusions
Description: Pericardial effusions: any pericardial effusion defined as at least moderate (i.e. measuring at least 2.0 cm in diastole, in the point of largest distance between the pericardial leaflets), with or without signs of hemodynamic compromise, or leading to drainage or to prolonged hospitalization. Pleural effusions: need for surgical drainage tubes for longer than 7 days after surgery and subsequent pleural effusions leading to drainage. CI = confidence interval, HR = hazard ratio, MDRD = Modification of Diet in Renal Disease
Time Frame: 6 months
Population: safety population
Measure: Number; unit: participants
Arm/Group | Immediate Introduction of Everolimus | Delayed Introduction of Everolimus
Number analyzed (Participants) | 89 | 87
participants | 30 | 18
Statistical Analysis 1: Comparison: Immediate Introduction of Everolimus vs Delayed Introduction of Everolimus; Test type: Superiority or Other; p = 0.0398, Regression, Cox; Hazard Ratio (HR) = 1.847, 95% CI 2-sided [1.029 to 3.315]

4. Secondary Outcome: Absolute and Percent Frequencies of Patients With LDL ≥ 100 mg/mL at 1, 3 and 6 Months, by Treatment Group
Description: LDL = low density lipoprotein
Time Frame: 6 months
Population: safety population
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Immediate Introduction of Everolimus | Delayed Introduction of Everolimus
Number analyzed (Participants) | 89 | 92
participants
  Month 1 | 41 [35.70 to 56.40] | 38 [31.60 to 51.90]
  Month 3 | 37 [32.60 to 53.50] | 37 [30.20 to 50.20]
  Month 6 | 34 [28.10 to 48.30] | 36 [29.20 to 49.10]

5. Secondary Outcome: Participants With CMV Infection and CMV Syndrome/Disease After 6 Months by Treatment Group
Description: CMV infection is defined as pp65 antigenemia or DNAemia
Time Frame: 6 months
Population: safety population
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Immediate Introduction of Everolimus | Delayed Introduction of Everolimus
Number analyzed (Participants) | 89 | 92
participants
  CMV infections | 46 [41.30 to 62.10] | 63 [59.00 to 78.00]
  CMV syndrome/disease | 3 [0.00 to 7.10] | 6 [1.50 to 11.60]
Statistical Analysis 1: Comparison: Immediate Introduction of Everolimus vs Delayed Introduction of Everolimus; CMV infections; Test type: Superiority or Other; p = 0.0234, Fisher Exact

6. Secondary Outcome: Participants With at Least One Occurrence of Composite Treatment Failure Events
Description: Comparison of 6-months cumulative incidence of composite treatment failure events (BPAR ≥ 2R, rejection with hemodynamic compromise, graft loss, or death) between delayed everolimus arm and immediate everolimus arm
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Immediate Introduction of Everolimus | Delayed Introduction of Everolimus
Number analyzed (Participants) | 89 | 92
participants | 33 [27.00 to 47.10] | 26 [19.10 to 37.50]
Statistical Analysis 1: Comparison: Immediate Introduction of Everolimus vs Delayed Introduction of Everolimus; Test type: Superiority or Other; p = 0.1966, Regression, Cox; Hazard Ratio (HR) = 1.403, 95% CI 2-sided [0.839 to 2.347]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Safety population
Arm/Group | Immediate Introduction of Everolimus | Delayed Introduction of Everolimus
Serious Adverse Events (participants affected / at risk) | 35/89 | 31/92
Other Adverse Events (participants affected / at risk) | 72/89 | 68/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Introduction of Everolimus (N=89) | Delayed Introduction of Everolimus (N=92)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 12 | 4
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Concomitant disease progression (General disorders) | 0 | 2
Death (General disorders) | 0 | 1
Drug interaction (General disorders) | 1 | 0
Hyperpyrexia (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 1
Sudden death (General disorders) | 1 | 0
Cholecystitis and cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Transplant rejection (Immune system disorders) | 7 | 3
Cytomegalovirus infection (Infections and infestations) | 4 | 6
Cytomegalovirus syndrome (Infections and infestations) | 0 | 3
Endocarditis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 2
Pyelonephritis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract infections (Infections and infestations) | 2 | 1
Incision site complication (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 3 | 1
Escherichia test positive (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic syndrome (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1
Femoral arterial stenosis (Vascular disorders) | 0 | 1
Femoral artery aneurysm (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Introduction of Everolimus (N=89) | Delayed Introduction of Everolimus (N=92)
Anaemia (Blood and lymphatic system disorders) | 9 | 9
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 16 | 7
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 4
Atrial fibrillation (Cardiac disorders) | 5 | 3
Atrial flutter (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Chest pain (Cardiac disorders) | 1 | 1
Dilatation ventricular (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 40 | 32
Sinus tachycardia (Cardiac disorders) | 3 | 4
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular hypokinesia (Cardiac disorders) | 0 | 1
Diabetes mellitus (Endocrine disorders) | 1 | 2
Hyperthyroidism (Endocrine disorders) | 1 | 1
Thyroid disorder (Endocrine disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Implant site haematoma (General disorders) | 1 | 0
Oedema (General disorders) | 4 | 1
Oedema peripheral (General disorders) | 5 | 3
Oedema perpheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 6
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 3
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Transplant rejection (Immune system disorders) | 28 | 23
Bronchitis (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 1 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 2 | 6
Epstein-Barr virus infection (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis aerobacter (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 2 | 2
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 5
Influenza (Infections and infestations) | 0 | 1
Mediastinitis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1
Oral stomatitis (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pseudomonal infectios (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Toxoplasmosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Urinary tract infections (Infections and infestations) | 6 | 3
Wound infection (Infections and infestations) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Sternal injury (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Tongue injury (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 8 | 8
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 1
Blood culture positive (Investigations) | 0 | 1
Blood iron decreased (Investigations) | 1 | 1
Blood potassium descreased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
CPK increase (Investigations) | 0 | 1
CSF white blood cell count increased (Investigations) | 0 | 1
Cytomegalovirus test positive (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 2 | 0
Muscle enzyme increased (Investigations) | 1 | 0
Platelet count descreased (Investigations) | 1 | 1
Red blood cell count decreased (Investigations) | 0 | 1
Transaminases (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2
Hyperlipidemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscoloskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 4 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 2
Spinal column injury (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon rupture (Musculoskeletal and connective tissue disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Hemianopia (Nervous system disorders) | 1 | 0
Hemicephalalgia (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Vertigo positional (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 0
Dysphoria (Psychiatric disorders) | 0 | 1
Fluid retention (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Hypercreatininaemia (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 5
Renal failure chronic (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 18 | 25
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory tract infecion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1
Transfusion (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Femoral artery aneurysm (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 10 | 11
Hypotension (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 3 | 0
Lymphocele (Vascular disorders) | 0 | 1
Polypoidal choroidal vasculopathy (Vascular disorders) | 0 | 1
Retinal vein thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.